CLINICAL TRIAL: NCT00413712
Title: Comparism Between Efficacy and Effectiveness Between Slow Infusion of Calcium Channel Blockers and Intravenous Bolus Adenosine in the Management of Supraventricular Tachycardia in the Emergency Department.
Brief Title: Effectiveness of Calcium Channel Blockers and Adenosine in the Emergency Management of SVT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB18/1997
Record Dates: First submitted 2006-12-19; First posted 2006-12-20 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Supraventricular Tachycardia
Keywords: Supraventricular Tachycardia; Calcium Channel Blockers; Verapamil; Diltiazem; Adenosine
MeSH Terms: conditions — Tachycardia, Supraventricular | interventions — Calcium Channel Blockers; Adenosine

INTERVENTIONS:
Drug: Calcium Channel Blocker & Adenosine

SUMMARY:
The purpose of this study is to determine the efficacy and effectiveness of calcium channel blockers and adenosine in the treatment of Supraventricular Tachycardia.

DETAILED DESCRIPTION:
Paroxysmal Supraventricular Tachycardia (SVT) is a common cardiac emergency encountered in the Emergency Department. Both Calcium Channel Blockers (CCB) and Adenosine have been using in the Management of SVT.

Objective

This study compared the efficacy and effectiveness between slow Infusion of Calcium Channel Blockers (either Verapamil or Diltiazem) and bolus intravenous Adenosine in termination of SVT.

Methodology

This was a prospective, randomised, controlled clinical trial comparing the efficacy and effects of intravenous adenosine with slow infusion of calcium channel blockers (verapamil or diltiazem) in patients presenting with SVT to an Emergency Department. The study was approved by the hospital's Ethics Committee.

Patients of at least 10 years of age, who presented to the Emergency Department of the Singapore General Hospital with regular narrow complex tachycardia and an electrocardiographic(ECG) diagnosis of SVT that was not converted by vagal manoeuvres (Valsava manoeuvre or carotid sinus massage or both) and who were in SVT at the time of doctor attendance were included in the study.

The exclusion criteria were as follows:

* Patients with signs of impaired cerebral perfusion (e.g. altered mental state) or acute pulmonary oedema
* Patients with a subsequent diagnosis of arrhythmias other than SVT (i.e. sinus tachycardia, atrial flutter, atrial fibrillation or idiopathic ventricular tachycardia) were excluded from the analysis if they were initially enrolled
* Pregnancy by history (urine pregnancy testing was not used to actively exclude the condition in any of the female patients entered into the study).

Having selected the patients according to the criteria, they were randomly assigned into two groups: one to receive calcium channel blockers and the other, Adenosine. Within the former group, some were assigned randomly to receive Diltiazem and some to Verapamil.

Diltiazem was given at the dose of 2.5mg per minute (4ml per minute of a concentration of 0.625 mg/ml) up to a maximum of 50 mg. The dose of Verapamil was 1mg per minute (4ml per minute of a concentration of 0.25mg/ml) up to a maximum of 20mg. Both were given as a slow intravenous infusion using a Terumo infusion pump.

During intravenous infusion, the patient's vital signs, viz. heart rate and systolic and diastolic blood pressures, were monitored at two-minute intervals up to completion of infusion or conversion from SVT, whichever was the earlier. At the time of conversion to sinus rhythm, the infusion was stopped and the amount of drug infused was noted and recorded.

Regarding the Adenosine group, all the patients were administered Adenosine as a rapid bolus within 2 sec through an 18G IV cannula at an antecubital vein, followed by 10 ml saline flush and elevation of the limb. Initially 6ml bolus was given rapidly, and if there was no conversion of the SVT within 2 min, another 12 mg bolus was administered.

If SVT was not converted at the end of any of calcium channel blocker infusion, those patients were then given intravenous Adenosine as described above. Similarly, those patients who remained in SVT after first two initial boluses of Adenosine were again randomized to receive either Verapamil or Diltiazem.

This allowed four orders of treatment as follows:

* Verapamil infusion followed by Adenosine
* Diltiazem infusion followed by Adenosine
* Adenosine followed by Verapamil infusion
* Adenosine followed by Diltiazem infusion

If the tachycardia was not converted at the end of the study protocol, patients were managed either with synchronised electrical cardioversion if haemodynamically unstable or with further pharmacotherapy at the discretion of the treating physician if vital signs were stable.

Following the successful conversion, patients' vital signs were closely monitored at 1 min (immediate post-conversion), 5,10, 15 min and finally 30 min of post-conversion. If they remained stable, they were shifted to observation ward with continuous telemetric monitoring. They were eventually discharged if there were no recurrence during the period of observation and arranged a follow-up appointment at Arrhythmia Clinic one week later. Patients with the recurrence of SVT during the two-hour observation period were managed at the discretion of the treating physician.

Study end points were as follows:

* Conversion to sinus rhythm
* Withdrawal because of major adverse effects
* Completion of trial protocol without termination of tachycardia

Data on the final analysis was obtained from follow-up records of Cardiology department as well. The cost of medication used for each patient was also computed to understand the cost aspects of different regimens.

ELIGIBILITY:
Inclusion Criteria:

* More than 10 years old
* Electrocardiographic diagnosis of SVT
* SVT not converted by the vagal manoeuvres

Exclusion Criteria:

* Signs of impaired cerebral perfusion
* Signs of pulmonary oedema
* Subsequent diagnosis of other types of arrythmias rather than SVT
* pregnancy by history

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 206
Dates: Start 1997-01; Study Completion 2001-03

PRIMARY OUTCOMES:
Conversion to the sinus rhythm.

SECONDARY OUTCOMES:
Recurrence of SVT
Stability of vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Lim S Han, MBBS,FRCS, Principal Investigator — Department of Emergency Medicine, Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

REFERENCES:
- [Background] Lim SH, Anantharaman V, Teo WS. Slow-infusion of calcium channel blockers in the emergency management of supraventricular tachycardia. Resuscitation. 2002 Feb;52(2):167-74. doi: 10.1016/s0300-9572(01)00459-2. PMID 11841884
- [Background] Brady WJ Jr, DeBehnke DJ, Wickman LL, Lindbeck G. Treatment of out-of-hospital supraventricular tachycardia: adenosine vs verapamil. Acad Emerg Med. 1996 Jun;3(6):574-85. doi: 10.1111/j.1553-2712.1996.tb03467.x. PMID 8727628
- [Background] Madsen CD, Pointer JE, Lynch TG. A comparison of adenosine and verapamil for the treatment of supraventricular tachycardia in the prehospital setting. Ann Emerg Med. 1995 May;25(5):649-55. doi: 10.1016/s0196-0644(95)70179-6. PMID 7741343
- [Background] Sethi KK, Singh B, Kalra GS, Arora R, Khalilullah M. Comparative clinical and electrophysiologic effects of adenosine and verapamil on termination of paroxysmal supraventricular tachycardia. Indian Heart J. 1994 May-Jun;46(3):141-4. PMID 7821934
- [Background] Viskin S, Belhassen B. Acute management of paroxysmal atrioventricular junctional reentrant supraventricular tachycardia: pharmacologic strategies. Am Heart J. 1990 Jul;120(1):180-8. doi: 10.1016/0002-8703(90)90176-x. PMID 2193494
- [Background] Camm AJ, Garratt CJ. Adenosine and supraventricular tachycardia. N Engl J Med. 1991 Dec 5;325(23):1621-9. doi: 10.1056/NEJM199112053252306. No abstract available. PMID 1944450
- [Background] Cairns CB, Niemann JT. Intravenous adenosine in the emergency department management of paroxysmal supraventricular tachycardia. Ann Emerg Med. 1991 Jul;20(7):717-21. doi: 10.1016/s0196-0644(05)80829-7. PMID 2064090
- [Background] DiMarco JP, Miles W, Akhtar M, Milstein S, Sharma AD, Platia E, McGovern B, Scheinman MM, Govier WC. Adenosine for paroxysmal supraventricular tachycardia: dose ranging and comparison with verapamil. Assessment in placebo-controlled, multicenter trials. The Adenosine for PSVT Study Group. Ann Intern Med. 1990 Jul 15;113(2):104-10. doi: 10.7326/0003-4819-113-2-104. PMID 2193560
- [Background] Belardinelli L, Linden J, Berne RM. The cardiac effects of adenosine. Prog Cardiovasc Dis. 1989 Jul-Aug;32(1):73-97. doi: 10.1016/0033-0620(89)90015-7. No abstract available. PMID 2664879
- [Background] Garratt C, Linker N, Griffith M, Ward D, Camm AJ. Comparison of adenosine and verapamil for termination of paroxysmal junctional tachycardia. Am J Cardiol. 1989 Dec 1;64(19):1310-6. doi: 10.1016/0002-9149(89)90573-0. PMID 2589197
- [Background] Belhassen B, Glick A, Laniado S. Comparative clinical and electrophysiologic effects of adenosine triphosphate and verapamil on paroxysmal reciprocating junctional tachycardia. Circulation. 1988 Apr;77(4):795-805. doi: 10.1161/01.cir.77.4.795. PMID 3349581
- [Background] Klein HO, Ninio R, Oren V, Lang R, Sareli P, DiSegni E, David D, Guerrero J, Kaplinsky E. The acute hemodynamic effects of intravenous verapamil in coronary artery disease. Assessment by equilibrium-gated radionuclide ventriculography. Circulation. 1983 Jan;67(1):101-10. doi: 10.1161/01.cir.67.1.101. PMID 6291805
- [Background] Betriu A, Chaitman BR, Bourassa MG, Brevers G, Scholl JM, Bruneau P, Gagne P, Chabot M. Beneficial effect of intravenous diltiazem in the acute management of paroxysmal supraventricular tachyarrhythmias. Circulation. 1983 Jan;67(1):88-94. doi: 10.1161/01.cir.67.1.88. PMID 6847809
- [Background] Mitchell LB, Schroeder JS, Mason JW. Comparative clinical electrophysiologic effects of diltiazem, verapamil and nifedipine: a review. Am J Cardiol. 1982 Feb 18;49(3):629-35. doi: 10.1016/s0002-9149(82)80022-2. PMID 6277182
- [Background] Singh BN, Hecht HS, Nademanee K, Chew CY. Electrophysiologic and hemodynamic effects of slow-channel blocking drugs. Prog Cardiovasc Dis. 1982 Sep-Oct;25(2):103-32. doi: 10.1016/0033-0620(82)90023-8. No abstract available. PMID 7051136
- [Background] Kawai C, Konishi T, Matsuyama E, Okazaki H. Comparative effects of three calcium antagonists, diltiazem, verapamil and nifedipine, on the sinoatrial and atrioventricular nodes. Experimental and clinical studies. Circulation. 1981 May;63(5):1035-42. doi: 10.1161/01.cir.63.5.1035. PMID 7471362
- [Background] Henderson AH, Lewis MJ. Basic mechanisms of 'calcium antagonists' (slow channel blockers). Scott Med J. 1981 Apr;26(2):156-60. doi: 10.1177/003693308102600215. No abstract available. PMID 6270785
- [Background] Russell DC. Electrophysiology and antiarrhythmic effects of calcium antagonists. Scott Med J. 1981 Apr;26(2):161-4. doi: 10.1177/003693308102600216. No abstract available. PMID 6270786
- [Background] Sung RJ, Elser B, McAllister RG Jr. Intravenous verapamil for termination of re-entrant supraventricular tachycardias: intracardiac studies correlated with plasma verapamil concentrations. Ann Intern Med. 1980 Nov;93(5):682-9. doi: 10.7326/0003-4819-93-5-682. PMID 7212475
- [Background] Seipel L, Breithardt G, Abendroth RR, Wiebringhaus E. [The electrophysiological effects of the Ca-antagonists gallopamil (D 600), dimeditiapramine (Ro 11-1781) and verapamil in man (author's transl)]. Z Kardiol. 1980 Aug;69(8):551-5. German. PMID 7445655
- [Background] Singh BN, Roche AH. Effects of intravenous verapamil on hemodynamics in patients with heart disease. Am Heart J. 1977 Nov;94(5):593-9. doi: 10.1016/s0002-8703(77)80128-2. PMID 333889
- [Background] Heng MK, Singh BN, Roche AH, Norris RM, Mercer CJ. Effects of intravenous verapamil on cardiac arrhythmias and on the electrocardiogram. Am Heart J. 1975 Oct;90(4):487-98. doi: 10.1016/0002-8703(75)90431-7. PMID 1163442
- [Background] Schamroth L, Krikler DM, Garrett C. Immediate effects of intravenous verapamil in cardiac arrhythmias. Br Med J. 1972 Mar 11;1(5801):660-2. doi: 10.1136/bmj.1.5801.660. PMID 5015294